CLINICAL TRIAL: NCT05370794
Title: Is in Vitro Maturation of Oocytes Influenced by the Origin of Gonadotropins Used in Maturation Medium: is There a Difference in Efficiency When Using Urinary Versus Recombinant Produced Follicle Stimulating Hormone and Human Chorionic Gonadotropin
Acronym: IVM-FSHhCG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-IVM-FSHhCG
Record Dates: First submitted 2022-04-04; First posted 2022-05-12 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-05

CONDITIONS: In Vitro Maturation of Oocytes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — spent medium after IVM, cumulus cells after IVM
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard IVM: urinary purified gonadotropins (uFSH and uhCG): uhCG = Pregnyl®, 5000IU/ vial, Organon-Merck: final concentration 100mIU/ml + uFSH = Menopur® 75mIU/ml, Ferring: final concentration 75mIU/ml.
  Administered during 30h of in vitro maturation culture
- Experimental IVM: recombinant gonadotropins (rFSH and rhCG): rhCG= Ovitrelle®, 250g/0.5ml = 26000IU/ml, Merck-Serono : final concentration 100mIU/ml + rFSH = Gonal F®, 300IU/0.5ml, Merck-Serono: final concentration 75mIU/ml.
  Administered during 30h of in vitro maturation culture
  Interventions: Drug: rhCG= Ovitrelle®, 250g/0.5ml = 26000IU/ml, Merck-Serono; Drug: rFSH = Gonal F®, 300IU/0.5ml, Merck-Serono

INTERVENTIONS:
Drug: rhCG= Ovitrelle®, 250g/0.5ml = 26000IU/ml, Merck-Serono — recombinant hCG
  Groups: Experimental IVM: recombinant gonadotropins (rFSH and rhCG)
Drug: rFSH = Gonal F®, 300IU/0.5ml, Merck-Serono — recombinant FSH
  Groups: Experimental IVM: recombinant gonadotropins (rFSH and rhCG)

SUMMARY:
Standard IVM currently contains urinary purified hormones which might contain contaminants possibly affecting maturation of embryo development. The investigators will test if the efficiency in terms of oocyte maturation after IVM of recombinant (without contaminants) is equivalent to urinary gonadotropins. Urinary and recombinant FSH and hCG will be used in equivalent bioactivity as measured in IU/ml and specified by the manufacturer. Sibling oocytes of the patient will be subjected to IVM medium containing urinary or recombinant gonadotropins. Oocyte maturation is the primary outcome, however, fertilization rate and preimplantation embryo development will be investigated.

DETAILED DESCRIPTION:
In vitro maturation is a valid option for PCO(S) patients in the daily ART clinic, however maturation and embryologic development are not yet matching the efficiency levels obtained by standard COS treatment (Ho et al. 2019). To further enhance embryo quality after IVM, media and supplements should be efficient, safe and pure. It has been described that a threshold of FSH activity is necessary for maturation in human IVM (Cadenas et al. 2021), but hCG might be redundant (Ge et al 2008).

Until now, the investigators have been using highly purified urinary derived gonadotropins to supplement IVM media. However in the last decades more recombinant products are available and thoroughly characterized. In ART, both urinary derived and recombinant produced hormones are used to induce multiple follicle growth and ovulation in an ovarian stimulation cycle. Due to the fear of transmis-sion of pathogens (though not yet documented) and of intolerance caused by contaminants, recombinant products are often preferred in the clinic, with no indications of differences in effectiveness and safety (Nahuis 2009). In an in vitro bioassay, contaminating proteins may alter biological re-sponses with undesired effects. uFSH is documented to contain e.g. Insulin-like growth factor binding protein 1 (IGFBP7), that may inhibit oestrogen production, and Eosinophil Derived Neurotoxin (EDN), with known inhibitory effects on mouse oocyte maturation (Bassett 2009). Hence it is important in an in vitro system to use products with the highest purity available.

Moreover the oligosaccharide sialylation is different depending on the production method, altering the acidity and hereby the half-life in the body, but more importantly for an in vitro system, also the receptor binding potency (Bassett 2009, Riccetti 2017).

Hence, before changing our standard system for a theoretically better alternative, The investigators need to test the efficiency of recombinant hormones compared to the routinely used urinary hormones in terms of oocyte maturation efficiency in the in vitro maturation system.

PCOS patients eligible for an IVM cycle to treat infertility will be included. Patients will receive a mild ovarian stimulation protocol, identical to our standard IVM care program.

The investigators will conduct a non-inferiority study for oocyte maturation efficiency with a limit of 10%, significance level of 5% and power of 80%, leading to a sample size of 618 oocytes. The investigators estimate this will be obtained if 35 patients are included in the study.

After OR follicle fluids containing COC are filtered over a 70µm mesh filter to eliminate contaminating blood cells and hereby visualizing the COC. The first detected COC will be transferred into a wash droplet of a 4-well dish, the second COC will be kept in the second wash droplet of the 4-well dish, … According to the randomization list, the COC in the first droplet of the 4-well dish will be allocated to the standard or experimental IVM. The randomization list is generated with www.sealedenvelope.com.

Mature oocytes will be ferilized by Intracytoplasmic Sperm Injection (ICSI) and fertilization and embryological development will be recorded. Embryos of sufficient quality on day 3 will be vitrified for a deferred vitrified/warmed embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* PCO(S) patients
* Anti-Mullerian Hormone ≥ 3.6 ng/mL
* Basal Antral Follicle Count ≥ 20
* All ranks of trial

Exclusion Criteria:

* Surgically obtained semen sample
* Grade 3 or 4 endometriosis, minor or major uterine abnormalities
* Preimplantation Genetic Testing
* Priming with Letrozole

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: infertility patients
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
oocyte maturation | oocyte maturation is assessed after 30 hours of in vitro maturation
  the ability of the oocyte to extrude the first polar body

SECONDARY OUTCOMES:
Fertilization rate | the presence of 2 pronuclei is assessed between 18-20 hours after ICSI
  the ability of the oocyte to ba activated and form pronuclei
morphologic parameters describing embryo quality per fertilized oocyte | embryo developmental assessment is performed 3 days after ICSI
  embryo developmental potential as estimated by morphological characteristics: embryos with 6 cells or more, less than 20% fragmentation, cell size according to division pattern and the absence of multinucleated blastomeres are considered as good quality embryos. As secondary parameters, the presence of vacuoles or granulation in the majority of blastomeres will exclude the embryo from the 'good quality' group regardless of the earlier mentioned parameters.
utilization rate | utilization rate will be established 3 days after ICSI
  the embryos of sufficient quality to be vitrified for a deferred embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Michel De Vos, MD,PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho VNA, Braam SC, Pham TD, Mol BW, Vuong LN. The effectiveness and safety of in vitro maturation of oocytes versus in vitro fertilization in women with a high antral follicle count. Hum Reprod. 2019 Jun 4;34(6):1055-1064. doi: 10.1093/humrep/dez060. PMID 31111879
- [Background] Cadenas J, Nikiforov D, Pors SE, Zuniga LA, Wakimoto Y, Ghezelayagh Z, Mamsen LS, Kristensen SG, Andersen CY. A threshold concentration of FSH is needed during IVM of ex vivo collected human oocytes. J Assist Reprod Genet. 2021 Jun;38(6):1341-1348. doi: 10.1007/s10815-021-02244-8. Epub 2021 May 28. PMID 34050448
- [Background] Ge HS, Huang XF, Zhang W, Zhao JZ, Lin JJ, Zhou W. Exposure to human chorionic gonadotropin during in vitro maturation does not improve the maturation rate and developmental potential of immature oocytes from patients with polycystic ovary syndrome. Fertil Steril. 2008 Jan;89(1):98-103. doi: 10.1016/j.fertnstert.2007.02.021. Epub 2007 May 24. PMID 17524398
- [Background] Nahuis M, van der Veen F, Oosterhuis J, Mol BW, Hompes P, van Wely M. Review of the safety, efficacy, costs and patient acceptability of recombinant follicle-stimulating hormone for injection in assisting ovulation induction in infertile women. Int J Womens Health. 2010 Aug 9;1:205-11. doi: 10.2147/ijwh.s4729. PMID 21072289
- [Background] Bassett R, Lispi M, Ceccarelli D, Grimaldi L, Mancinelli M, Martelli F, Van Dorsselaer A. Analytical identification of additional impurities in urinary-derived gonadotrophins. Reprod Biomed Online. 2009 Sep;19(3):300-13. doi: 10.1016/s1472-6483(10)60163-0. PMID 19778474
- [Background] Riccetti L, Klett D, Ayoub MA, Boulo T, Pignatti E, Tagliavini S, Varani M, Trenti T, Nicoli A, Capodanno F, La Sala GB, Reiter E, Simoni M, Casarini L. Heterogeneous hCG and hMG commercial preparations result in different intracellular signalling but induce a similar long-term progesterone response in vitro. Mol Hum Reprod. 2017 Oct 1;23(10):685-697. doi: 10.1093/molehr/gax047. PMID 29044421